CLINICAL TRIAL: NCT03031925
Title: Detection of Annexin A2 in Systemic Lupus Erythematosus
Acronym: ANLUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI2017_843_0001
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis
Keywords: Annexin A2; biomarker
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLE patients (Experimental): Systemic Lupus Erythematosus
  Interventions: Other: ANXA2
- control subjects (Active Comparator): age- and sex-matched control subjects
  Interventions: Other: ANXA2

INTERVENTIONS:
Other: ANXA2 — serum and urinary concentration

SUMMARY:
There is substantial clinical and biological intra and inter-patient variability in SLE. Vascular, renal and neurologic deficiency can be organ-threatening or even life-threatening, leading to increased morbidity and mortality.

Thus, biomarkers of disease activity and prognosis are required for regular follow-up of SLE patients.

Implication of Toll-like Receptors (TLRs) in SLE has been extensively studied in mice models and humans. Self nuclear antigens bind to TLRs which are located on the surface of dendritic cells, B-cells, and endothelial cells, leading to production of pro-inflammatory cytokines and pathologic autoantibodies involved in organ dysfunction of SLE patients. Moreover, TLR expression in SLE is significantly higher and significantly correlated with disease activity.

Annexin A2 (ANXA2) is a member of the annexins superfamily which exists as a monomer or heterotetramer and is implicated in several biological processes. Most notably, it binds to ẞ2GP1/anti-ẞ2GP1 antibodies and mediates endothelial cell activation via a TLR4 signaling pathway, highlighting its key role in Antiphospholipid Syndrome (APS) frequently associated with SLE.

ANXA2 is also involved in the physiopathology of SLE. Anti-DNA autoantibodies can bind with ANXA2 expressed on mesangial cells in lupus nephritis. Besides, a french study carried out in Amiens' University Hospital showed that vascular lesions in lupus nephritis were associated with a significant increase in vascular expression of ANXA2.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients :

* Age ≥ 18 years old
* All SLE patients fulfilling the 1997 ACR criteria, followed at the Departments of Internal Medicine and Nephrology at CHU Amiens-Picardie, regardless of clinical status, treatment, and disease activity.
* Written informed consent

Inclusion criteria for control subjects :

* Age ≥ 18 years old
* Written informed consent

The patients will be compared with age- and sex-matched control subjects.

Exclusion Criteria:

* drug-induced lupus erythematosus
* refusal or incapacity to provide a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
serum concentration of ANXA2 | Day 0
urinary concentration of ANXA2 | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Valéry SALLE, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France